CLINICAL TRIAL: NCT00090727
Title: A Phase 1, Open-Label, Dose-Escalation Study of AQ4N Administered Intravenously in Patients With Advanced Malignancies
Brief Title: Chemotherapy for Patients With Advanced Solid Tumors or Non-Hodgkin's Lymphoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Novacea (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 021-001
Record Dates: First submitted 2004-09-02; First posted 2004-09-06 (Estimated); Last update posted 2006-11-02 (Estimated); Status verified 2005-04

CONDITIONS: Solid Malignancies; Non-Hodgkin's Lymphoma
Keywords: diffuse; follicular; chronic lymphocytic leukemia; colorectal cancer; pancreatic cancer; acute myelogenous leukemia; head and neck cancer; breast cancer; prostate cancer; ovarian cancer; bladder cancer; hypoxia; refractory; metastatic
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Leukemia, Lymphocytic, Chronic, B-Cell; Colorectal Neoplasms; Pancreatic Neoplasms; Leukemia, Myeloid, Acute; Head and Neck Neoplasms; Breast Neoplasms; Prostatic Neoplasms; Ovarian Neoplasms; Urinary Bladder Neoplasms; Hypoxia; Neoplasm Metastasis | interventions — AQ4N

INTERVENTIONS:
Drug: AQ4N

SUMMARY:
The purposes of this study are to determine:

* the largest dose of AQ4N that can be safely given once a week for three weeks out of a 4 week cycle
* the side effects of AQ4N when given on the above schedule
* how much AQ4N is in the blood and urine at specific times after administration and how the body get rids of AQ4N
* if AQ4N helps treat cancer

DETAILED DESCRIPTION:
This study is for people who have advanced cancer for which standard chemotherapy did not work or for which there are no reliably, effective treatments.

AQ4N is an experimental chemotherapy that is thought to target tumor areas with low oxygen content and low blood supply; tumor areas that are usually the most resistant to standard chemotherapy and radiation treatment. AQ4N may be beneficial in cancer treatment by interfering with a protein that is required for cells to grow and divide, causing tumors to die or to delay their growth.

All patients in this study will receive AQ4N. The dose will be increased for each new patient or group of patients until the maximum tolerated dose is reached.

ELIGIBILITY:
Inclusion Criteria:

* Advanced solid malignancy or non-Hodgkin's lymphoma that is refractory to treatment or has recurred
* Age > 18 years
* Adequate hematologic (blood), kidney and liver function
* Negative pregnancy test (females of childbearing potential only)
* Willingness to use effective contraception by both males and females throughout the treatment period and for at least 2 months following treatment.

Exclusion Criteria:

* Any chemotherapy or radiation within the past 4 weeks
* Symptomatic or uncontrolled brain metastases (patients with history of brain metastases who have had repeat brain scans within the past 30 days that demonstrate no evidence of tumor progression or brain swelling and who do not require corticosteriod treatment may be eligible)
* Significant cardiovascular illness including, but not limited to, the following: active infection, uncontrolled hypertension, symptomatic congestive heart failure, unstable angina pectoris, heart attack within the past six months, or uncontrolled, irregular heart beat
* Inadequate cardiac function
* Prior investigational therapy within the past 28 days
* Pregnant or breast feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45
Dates: Start 2004-08

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Weiler Hospital of Albert Einstein College of Medicine, The Bronx, New York
  - Cancer Therapy & Research Center / Institute for Drug Development, San Antonio, Texas